CLINICAL TRIAL: NCT04033419
Title: Memantine for Prevention of Cognitive Decline During Adjuvant or Neoadjuvant Chemotherapy in Patients With Breast Cancer
Brief Title: Memantine for Prevention of Cognitive Decline in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LCCC1921; 5K12HD001441 (NIH)
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Decline; Chemo-brain
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Memantine (Experimental): Subjects receive memantin
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — memantine dose
  * Week 1: 5 mg dose once daily
  * Week 2: 5 mg dose twice daily
  * Week 3: 5 mg each morning/10 mg each evening
  * Week 4 through the end of Chemotherapy: 10 mg dose twice daily
  * Total duration: 12 - 26 weeks (depending on chemotherapy regimen)
  Other Names: Namenda

SUMMARY:
Purpose: To conduct a one-arm phase II trial to: (1) compare changes in pre- to post-chemotherapy cognitive function in a cohort of patients with breast cancer receiving memantine to historical controls; (2) examine how depression, anxiety, fatigue, baseline Intelligence Quotient (IQ), and cognitive effort relate to objective and self-reported cognitive function; and (3) estimate the feasibility of conducting a clinical trial of memantine for attenuating cognitive decline in patients with breast cancer during chemotherapy.

Participants: Adult patients with stage I-III breast cancer scheduled for adjuvant or neoadjuvant chemotherapy.

Procedures (methods): Cognitive assessments will be performed within one week of initiating and four weeks after completion of chemotherapy. Patients will receive memantine 10 mg twice daily between the pre- and post-chemotherapy study assessments. Cognitive function will be assessed objectively using a computerized cognitive test (Delayed Matching to Sample (DMS) test) and a standard neuropsychological battery. To assess subjective cognitive function, the Patient Reported Outcome Measurement Information System (PROMIS) Cognitive Function measure will be used. Depression, anxiety, fatigue, menopausal status, and sleep will be assessed as covariates.

DETAILED DESCRIPTION:
This is a one-arm phase II interventional study in patients with breast cancer to investigate whether memantine can prevent cognitive decline during chemotherapy. The investigators will recruit 56 participants referred to the University of North Carolina (UNC) Breast Center and affiliated outpatient clinics for initiation of adjuvant or neoadjuvant chemotherapy, perform a cognitive assessment within one week of initiating and four weeks after completion of chemotherapy, and treat with memantine 10 mg twice daily between the pre- and post-chemotherapy study assessments (estimated duration: 12-26 weeks, depending on the chemotherapy regimen). Cognitive function will be assessed objectively using a computerized cognitive assessment (Delayed Matching to Sample (DMS) test) and a standard neuropsychological battery. To assess subjective cognitive function, the Patient Reported Outcome Measurement Information System (PROMIS) Cognitive Function measure will be used. Depression, anxiety, fatigue, menopausal status, and sleep are comorbidities known to affect cognitive function, and therefore will be assessed as covariates pre- and post-chemotherapy. Depression, anxiety, health-related quality of life (HRQOL) and functional status will be evaluated as secondary outcomes. The feasibility of the investigator's study by monitoring recruitment, retention, and adherence to memantine will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* At least 18 years of age
* Able to speak English
* Diagnosed with breast cancer, Stages I-III
* Scheduled for adjuvant or neoadjuvant chemotherapy

Exclusion Criteria:

* A history of adverse reaction to memantine
* Another cancer diagnosis with an estimated survival of less than five years
* Previous chemotherapy exposure
* Severe cognitive impairment, defined as Blessed Orientation Memory Concentration Test (BOMC) ≥ 11.
* Pregnancy, confirmed by a negative pregnancy test within 30 days of study enrollment, or breastfeeding
* Current alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zev M Nakamura, MD, Principal Investigator — Univesity of North Carolina at Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: IRB, IEC, or REB approval, as applicable, and execution of a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Nakamura ZM, Deal AM, Park EM, Stanton KE, Lopez YE, Quillen LJ, O'Hare Kelly E, Heiling HM, Nyrop KA, Ray EM, Dees EC, Reeder-Hayes KE, Jolly TA, Carey LA, Abdou Y, Olajide OA, Rauch JK, Joseph R, Copeland A, McNamara MA, Ahles TA, Muss HB. A phase II single-arm trial of memantine for prevention of cognitive decline during chemotherapy in patients with early breast cancer: Feasibility, tolerability, acceptability, and preliminary effects. Cancer Med. 2023 Apr;12(7):8172-8183. doi: 10.1002/cam4.5619. Epub 2023 Jan 16. PMID 36645168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 09/25/2019 through 08/13/2021 at six cancer centers in North Carolina.
Pre-assignment Details: A total of fifty-six participants consented to the study, but one of them was deemed to be ineligible therefore 55 participants were enrolled in the study.
Groups:
- Memantine: Memantine: - Week 1: 5 mg dose once daily
  * Week 2: 5 mg dose twice daily
  * Week 3: 5 mg each morning/10 mg each evening
  * Week 4 through end of Chemotherapy: 10 mg dose twice daily
  * Total duration: 12 - 26 weeks (depending on chemotherapy regimen)
Period: Overall Study
Arm/Group | Memantine
Started | 51
Completed | 45
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants
Arm/Group | Memantine
Number analyzed (Participants) | 55
Age, Continuous [Mean (Full Range); unit: years] | 56.1 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 42
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Working Memory - Delayed Matching to Sample Test
Description: The Delayed Matching to Sample Test (DMS) is a computerized cognitive assessment of visual working memory. The DMS will be administered using Cambridge Neuropsychological Test Automated Battery (CANTAB) eclipse software (Cambridge Cognition, Cambridge, UK). The participant is shown an image with four patterns and asked to match patterns simultaneously or after delay. The investigators will use the percent correct (0 to 100, higher is better) at the 12-second delay on the DMS test for the primary analysis.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: Forty-five subjects had at least one dose of memantine and completed both pre- and post-assessments and, thus, were evaluable for cognitive change.
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: Subjects received memantine and completed the visual working memory - Delayed Matching to Sample Test
Arm/Group | Memantine
Number analyzed (Participants) | 45
Participants
  Improved | 16
  No Change | 13
  Declined | 16

2. Secondary Outcome: Change in Verbal Memory - Hopkins Verbal Learning Test-Revised
Description: The Hopkins Verbal Learning Test-Revised (HVLT-R) is an objective measure of verbal learning and memory. The examiner reads a list of 12 nouns to the participant, who repeats as many words as remembered. Approximately 20-25 minutes later, participants are asked to recall as many words as possible. Then, the examiner reads a list of 24 words, including the 12 words from the original list, and the participant is asked to determine which words were and were not on the original list. These tasks result in three subscales: total recall (range: 0-36; higher is better), delayed recall (range: 0-12; higher is better), and the Recognition Discrimination Index (range: 0-12; higher is better).
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: Subjects received memantine and completed the HVLT-R test.
Arm/Group | Memantine
Number analyzed (Participants) | 45
Participants
  Improved | 22
  No Change | 16
  Declined | 7

3. Secondary Outcome: Change in Processing Speed and Executive Function - Trail Making Test
Description: The Trail Making Test (TMT) is an objective measure of processing speed (part A) and executive function (part B). In part A, the participant is given a diagram of 25 circles, labeled 1 - 25, and asked to connect the circles in ascending order. In part B, the diagram of 25 circles includes some with numbers (1-13) and some with letters (A-L), and the participant is asked to connect the circles alternating between numbers and letters. Performance is measured in the number of seconds required to complete each task (lower is better).
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: The participants received memantine and completed both pre- and post-assessments. Due COVID-19 pandemic, only 3 participants received memantine and completed both pre- and post-assessments. Their data was entered.
Measure: Mean (Standard Deviation); unit: time seconds
Groups:
- The Trail Making Test PART A Time (Secs.); The Trail Making Test PART B Time (Secs.): Participants received memantine and completed both pre- and post-assessments.
Arm/Group | The Trail Making Test PART A Time (Secs.) | The Trail Making Test PART B Time (Secs.)
Number analyzed (Participants) | 3 | 3
time seconds
  Baseline | 27.58 (2.325) | 79.42 (25.54)
  Post-chemotherapy | 32.65 (11.32) | 87.53 (11.32)

4. Secondary Outcome: Change in Processing Speed - Rapid Visual Processing (RVP)
Description: The Rapid Visual Processing test (RVP) is a computerized cognitive assessment of processing speed and sustained attention. The RVP will be administered using Cambridge Neuropsychological Test Automated Battery (CANTAB) eclipse software (Cambridge Cognition, Cambridge, UK). The participant is shown a series of pseudo-random digits from 2 to 9 and asked to recognize target digit sequences by pressing a button on the screen as quickly as possible. The investigators will measure total correct responses (higher is better).
  This test was added at the start of the COVID-19 pandemic as a substitute for the Trail Making Test.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: Forty-five subjects had at least one dose of memantine and completed both pre- and post-assessments. There are data available for 31 subjects.
  and, thus, were evaluable for cognitive change.
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: Subjects received memantine and completed The Rapid Visual Processing test (RVP) test
Arm/Group | Memantine
Number analyzed (Participants) | 31
Participants
  Improved | 10
  No Change | 17
  Declined | 4

5. Secondary Outcome: Change in Executive Function - One Touch Stockings (OTS) of Cambridge
Description: The One Touch Stockings (OTS) of Cambridge is a computerized cognitive assessment of executive function. The OTS will be administered using Cambridge Neuropsychological Test Automated Battery (CANTAB) eclipse software (Cambridge Cognition, Cambridge, UK). The participant is shown two displays with three colored balls presented as stacks suspended from a beam and a row of numbered boxes along the bottom of the screen. The participant is asked to work out in their head how many moves are required to match the two displays. The investigators will measure mean number of choices to the correct response (lower is better).
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: This test was added at the start of the COVID-19 pandemic as a substitute for the Trail Making Test. Accordingly, 31 subjects had at least one dose of memantine and completed both pre- and post-assessments and, thus, were evaluable for cognitive change.
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: Subjects received memantine and completed the One Touch Stockings (OTS) of Cambridge
Arm/Group | Memantine
Number analyzed (Participants) | 31
Participants
  Improved | 9
  No Change | 16
  Declined | 6

6. Secondary Outcome: Change in Attention and Working Memory - Digit Span
Description: The Digit Span is an objective measure of attention and working memory. The participant is asked to recite sequences of numbers in forward, backwards, and sequential order. The score for each sequence type is the number of correct responses (higher is better).
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: Subjects received memantine and completed the Digit Span test
Arm/Group | Memantine
Number analyzed (Participants) | 45
Participants
  Improved | 7
  No Change | 31
  Declined | 7

7. Secondary Outcome: Change in Verbal Fluency - Controlled Oral Word Association Test
Description: The Controlled Oral Word Association Test (COWA) is an objective measure of verbal fluency. The participant is asked to name as many words as possible, excluding proper nouns, in one minute. This is repeated for a total for three different letters. The score is the total number of different words produced between all three letters (higher is better).
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: The subjects received memantine and completed The Controlled Oral Word Association Test
Arm/Group | Memantine
Number analyzed (Participants) | 45
Participants
  Improved | 18
  No Change | 18
  Declined | 9

8. Secondary Outcome: Change in Semantic Fluency - Animal Naming Test
Description: The Animal Naming Test (ANT) is an objective measure of semantic fluency. The participant is asked to name as many animals as possible in one minute. The score is the number of unique animals stated (higher is better).
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: The subjects received memantine and completed The Animal Naming Test (ANT).
Arm/Group | Memantine
Number analyzed (Participants) | 45
Participants
  Improved | 10
  No Change | 16
  Declined | 19

9. Secondary Outcome: Change in Self-reported Cognitive Function - PROMIS Cognitive Function
Description: The National Institute of Health's Patient-Reported Outcomes Measurement Information System (PROMIS) contains a cognitive function bank. The PROMIS Cognitive Function 8a short form will be used. Scores for all PROMIS measures are reported on the T-score metric in which the mean=50 and standard deviation (SD) = 10 are centered on the general population means. Higher scores represent greater degrees of cognitive complaints.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: Forty-four subjects had at least one dose of memantine and completed both pre- and post-assessments and, thus, were evaluable for cognitive change.
Measure: Count of Participants; unit: Participants
Groups:
- Initial Normal Function; Initial Mild Decline; Initial Severe Decline: Baseline Cognitive Function based on PROMIS patient-reported outcome
Arm/Group | Initial Normal Function | Initial Mild Decline | Initial Severe Decline
Number analyzed (Participants) | 33 | 10 | 1
Participants
  Normal Function at Follow-Up | 18 | 2 | 1
  Decline to Mild at Follow-Up Cognitive Difficulties | 14 | 8 | 0
  Decline to Moderate at Follow-Up Cognitive Difficulties | 1 | 0 | 0

10. Secondary Outcome: Change in Depressive Symptoms - PROMIS Depression
Description: The National Institute of Health's Patient-Reported Outcomes Measurement Information System (PROMIS) contains a depression bank. The PROMIS Depression 8a short form will be used. Scores for all PROMIS measures are reported on the T-score metric in which the mean=50 and standard deviation (SD) = 10 are centered on the general population means. Higher scores represent greater degrees of depression. We evaluated the proportion of patients with at least moderately severe symptoms (T-score ≥ 65) at baseline and follow-up.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: Fifty-one subjects provided data regarding depression symptoms at baseline and forty-four provided data at follow-up. All available data were included to evaluate changes in depressive symptoms.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Depression: Subjects who had at least one dose of memantine and completed a baseline assessment of depression
- Post-assessment Depression: Subjects who had at least one dose of memantine and completed post-assessment of depression
Arm/Group | Baseline Depression | Post-assessment Depression
Number analyzed (Participants) | 51 | 44
Participants
  PROMIS Depression Score <65 | 50 | 43
  PROMIS Depression Score Value ≥ 65 | 1 | 1

11. Secondary Outcome: Change in Anxiety Symptoms - PROMIS Emotional Distress-Anxiety
Description: The National Institute of Health's Patient-Reported Outcomes Measurement Information System (PROMIS) contains an anxiety bank. The PROMIS Emotional Distress-Anxiety - Short Form 6a will be used. Scores for all PROMIS measures are reported on the T-score metric in which the mean=50 and standard deviation (SD) = 10 are centered on the general population means. Higher scores represent greater degrees of anxiety. We evaluated the proportion of patients with at least moderately severe symptoms (T-score ≥ 65) at baseline and follow-up.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy.
Population: Anxiety was assessed using the PROMIS Emotional Distress-Anxiety measure, in 51 subjects at baseline (all enrolled who had at least one dose of memantine) and in 45 subjects at the post-assessment (all who completed this measure at the post-assessment timepoint and had at least one dose of memantine)
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Anxiety: Subjects who had at least one dose of memantine and completed a baseline assessment of anxiety
- Post-assessment Anxiety: Subjects who had at least one dose of memantine and completed post-assessment of anxiety
Arm/Group | Baseline Anxiety | Post-assessment Anxiety
Number analyzed (Participants) | 51 | 45
Participants
  PROMIS Anxiety Score <65 | 48 | 40
  PROMIS Anxiety Score ≥ 65 | 3 | 5

12. Secondary Outcome: Change in Karnofsky Performance Status
Description: The number of subjects with Karnofsky Performance Status equal to or more than 80, at baseline and 4 weeks after chemotherapy were compared.
  The Patient-reported Karnofsky Performance Status (KPS) provides a self-characterization of functional status, ranging from severe/requiring continuous nursing care to normal/no complaints/no symptoms of the disease. Scores range from 30 to 100. Higher scores indicate better function.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: Karnofsky Performance Status of subjects was assessed both at baseline and 4 weeks after the completion of chemotherapy.
Measure: Count of Participants; unit: Participants
Groups:
- Karnofsky Performance Status Change: Karnofsky Performance Status of subjects was assessed both at baseline and 4 weeks after the completion of chemotherapy.
Arm/Group | Karnofsky Performance Status Change
Number analyzed (Participants) | 42
Participants
  Baseline Karnofsky Performance Status: => 80 | 37
  Baseline Karnofsky Performance Status: <80 | 5
  Post-treatment Karnofsky Performance Status: => 80 | 39
  Post-treatment Karnofsky Performance Status: <80 | 3

13. Secondary Outcome: Change in Quality of Life - Functional Assessment of Cancer Therapy-General
Description: The Functional Assessment of Cancer Therapy-General (FACT-G) is a 27-item patient-administered assessment of general quality-of-life measures in cancer patients. It has been validated in the literature and permits the measurement of a number of symptoms including nausea, pain, and insomnia. Responses to each item are on a 5-point Likert scale. The FACT-G total score (range: 0-108; higher is better) will be assessed.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: Subjects FACT-G scores were assessed both at baseline and 4 weeks after the completion of chemotherapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- FACT-G Scores Change: FACT-G scores of subjects was assessed both at baseline and 4 weeks after the completion of chemotherapy.
Arm/Group | FACT-G Scores Change
Number analyzed (Participants) | 43
score on a scale
  Baseline FACT-G | 83.7 (15.1)
  Post-treatment FACT-G | 82.6 (13.9)

14. Secondary Outcome: Proportion of Invited Participants Who Enroll - Recruitment
Description: Feasibility will be based on recruitment success as measured by the proportion of invited participants who enroll.
Time Frame: Baseline (pre-chemotherapy) over the duration of the accrual period
Population: The number of subjects who were assessed for eligibility enrolled and withdrawn.
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: The subjects who were invited to the study enrolled, received, and completed the treatment.
Arm/Group | Memantine
Number analyzed (Participants) | 412
Participants
  Assessed for eligibility | 412
  Enrolled | 55
  Withdrew | 4
  Received at least 1 dose | 51

15. Secondary Outcome: Proportion of Enrolled Participants Who do Not Meet the Primary Outcome Measure - Attrition
Description: Feasibility will be based on retention success as measured by the proportion of enrolled participants who are not eligible for analysis of the primary outcome.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: The subject received at least one dose of memantine.
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: 10 mg twice a day
Arm/Group | Memantine
Number analyzed (Participants) | 51
Participants
  Evaluable | 45
  Withdrew | 3
  Lost to follow-up | 3

16. Secondary Outcome: Proportion of Scheduled Drug Doses Taken - Adherence
Description: Feasibility will be based on adherence success as measured by the proportion of self-reported doses of memantine taken.
Time Frame: From baseline (pre-chemotherapy) to 4 weeks post-chemotherapy
Population: All subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: The subjects received memantine
Arm/Group | Memantine
Number analyzed (Participants) | 55
Participants
  never initiated memantine | 4
  >= 90% compliance | 39
  <90% compliance | 12

17. Secondary Outcome: Number of Adverse Events - Safety
Description: Safety is based on the number of all adverse events (AE) associated with memantine. The following most common side effects of memantine were explicitly solicited: headache, dizziness, confusion, constipation, diarrhea, and fatigue.
  AE was assessed and graded according to the NCI Common Terminology Criteria. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: From baseline to 4 weeks after chemotherapy (up to 30 weeks)
Population: All subjects who received at least one dose of memantine were assessed for adverse events. Four of the 55 subjects who enrolled did not receive memantine and were not evaluated for adverse events.
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: All subjects who received at least one dose of memantine were evaluated for adverse events.
Arm/Group | Memantine
Number analyzed (Participants) | 51
Participants
  fatigue | 19
  headache | 16
  constipation | 12
  diarrhea | 12
  dizziness | 10
  confusion | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from day one of the study drug administration to 4 weeks after completion of treatment (up to 30 weeks).
Description: AE were assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0. All patient-reported symptoms were recorded and examined for their association with memantine. Adverse Events associated with memantine. The most common adverse events of memantine: headache, dizziness, confusion, constipation, diarrhea, and fatigue were specifically collected.
Groups:
- All Subjects: Subjects who had at least one dose of memantine.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 40/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=51)
Anemia (Blood and lymphatic system disorders) | 4
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
blurred vision (Eye disorders) | 1
abdominal pain (Gastrointestinal disorders) | 2
constipation (Gastrointestinal disorders) | 12
diarrhea (Gastrointestinal disorders) | 12
dyspepsia (Gastrointestinal disorders) | 2
gastritis (Gastrointestinal disorders) | 1
gastrointestinal pain (Gastrointestinal disorders) | 1
gastrointestinal reflux (Gastrointestinal disorders) | 1
hematochezia (Gastrointestinal disorders) | 1
hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 7
vomiting (Gastrointestinal disorders) | 1
Chills (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 19
fever (General disorders) | 1
Generalized edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
lung infection (Infections and infestations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine Increased (Investigations) | 2
hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 3
hypocalcemia (Metabolism and nutrition disorders) | 2
hypokalemia (Metabolism and nutrition disorders) | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Cognitive disturbance (Nervous system disorders) | 5
confusion (Nervous system disorders) | 4
Depressed level of consciousness (Nervous system disorders) | 1
dizziness (Nervous system disorders) | 10
Extrapyramidal disorder (Nervous system disorders) | 1
headache (Nervous system disorders) | 16
Memory Impairment (Nervous system disorders) | 1
paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
insomnia (Psychiatric disorders) | 7
Restlessness (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
rash (pistular) (Skin and subcutaneous tissue disorders) | 7
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT04033419/Prot_SAP_000.pdf